CLINICAL TRIAL: NCT05941910
Title: The Effect of 6-month Treatment With Coenzyme Q10 on Endothelial, Vascular and Myocardial Function in Patients With Non-alcoholic Fatty Liver Disease
Brief Title: The Effect of Coenzyme Q10 on Endothelial, Vascular and Myocardial Function
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, VAIA LAMBADIARI, Professor of Internal Medicine-Endocrinology, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Q10nafldtrial
Record Dates: First submitted 2023-06-26; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Non-alcoholic fatty liver disease; endothelial function; vascular function; myocardial function; coronary flow reserve; endothelial glycocalyx; flow mediated dilation
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Tuberculin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Q10 (Active Comparator)
  Interventions: Drug: Q10
- Placebo (Placebo Comparator)
  Interventions: Drug: Q10

INTERVENTIONS:
Drug: Q10 — 240mg of Q10 orally, every day

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is associated with increased cardiovascular risk. The aim of this study is to investigate the effects of coenzyme Q10 (CoQ10) on endothelial, vascular and myocardial function in patients with NAFLD

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is associated with increased cardiovascular risk. The aim of this study is to investigate the effects of coenzyme Q10 (CoQ10) on endothelial, vascular and myocardial function in patients with NAFLD. In this trial patients with NAFLD will receive 240mg Q10 or placebo. At baseline and at 6 months, will be measured: a) Perfused boundary region (PBR) of the sublingual vessels using the SideviewDarkfieldimaging technique (Microscan, Glycocheck), b) pulse wave velocity (PWV-Complior, ALAM), c) flow-mediated dilation (FMD) of the brachial artery, d) left ventricular (LV) global longitudinal strain (GLS), and e) controlled attenuation parameter (CAP)for the quantification of liver steatosis by liver elastography (Fibroscan, Echosens).

ELIGIBILITY:
Inclusion Criteria:

* NAFLD AND one of below :

  1. dyslipidemia, as it is defined in the metabolic syndrome
  2. increased waist circumference as defined in the metabolic syndrome
  3. Arterial hypertension,
  4. overweight, (BMI>25)
  5. polycystic ovary syndrome,

Exclusion Criteria:

* Chronic Kidney Disease
* Heart Failure
* Liver failure
* Pregnancy/ Breast feeding
* Active malignancy (receiving Chemotherapy/immunotherapy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-08-14 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The effect of Q10 on Left Ventricular Myocardial Function | Six months
  The effect of Q10 on Left Ventricular Global Longitudinal Strain after six month administration of Q10

CONTACTS AND LOCATIONS:
Locations (1):
- Vaia Lambadiari, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vrentzos E, Ikonomidis I, Pavlidis G, Katogiannis K, Korakas E, Kountouri A, Pliouta L, Michalopoulou E, Pelekanou E, Boumpas D, Lambadiari V. Six-month supplementation with high dose coenzyme Q10 improves liver steatosis, endothelial, vascular and myocardial function in patients with metabolic-dysfunction associated steatotic liver disease: a randomized double-blind, placebo-controlled trial. Cardiovasc Diabetol. 2024 Jul 10;23(1):245. doi: 10.1186/s12933-024-02326-8. PMID 38987784